CLINICAL TRIAL: NCT04443738
Title: Long Term Follow up of Spinal Stenosis Inpatients Treated With Korean Integrative Medicine Treatment.
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2020-06
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Spinal Stenosis Lumbar; Medicine, Korean Traditional
Keywords: acupuncture therapy; herbal medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone survey — A questionnaire about the current symptoms and satisfaction for recieved treatment will be conducted over the phone for patients.

SUMMARY:
The purpose of this study is to reveal the effectiveness and safety of integrative Korean medicine for spinal stenosis by observation inpatients treated with integrative Korean medicine.

DETAILED DESCRIPTION:
This study is a prospective observational study. The subjects for study are patients diagnosed with spinal stenosis and who have been admitted to four Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, and Haeundae) for 2015.01-2018.12.

Medical records of selected patients will be analyzed, and telephone surveys will be conducted for each patient. The survey questions are Numeric rating scale (NRS), Oswestry disability index (ODI), quality of life, and Patient Global Impression of Change (PGIC), etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with spinal stenosis by an Korean medicine doctor and was admitted to Jaseng hospital of Korean medicien.
* Patients undergone MRI readings of central spinal stenosis
* Patients have no communication problems
* Patients have agreed to participate the study.

Exclusion Criteria:

* Patients who have been diagnosed with certain serious diseases that may cause back pain or neck pain (tumor metastases to the spine, acute fractures, spinal dislocations, and so on)
* Patient hospitalized for pain caused by a traffic accident
* Patients with serious mental illness
* Patients deemed unable to participate in the clinical research by other researchers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects for study are patients diagnosed with spinal stenosis and who have been admitted to four Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, and Haeundae) for 2015.01-2018.12.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | Finish survey by August 2020
  NRS uses an 11-point scale to evaluate current neck pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'. NRS was assessed at admission, 2 weeks after admission, discharge, and long term follow up.

SECONDARY OUTCOMES:
Oswestry disability index (ODI) | Finish survey by August 2020
  he ODI is a 10-item questionnaire developed to evaluate the degree of disability for low back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. We will conduct an validated Korean ODI questionnaire
The five level version of EuroQol-5 Dimension (EQ-5D) | Finish survey by August 2020
  EQ-5D is most widely used as a method of indirectly calculating the quality of life from various aspects. The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about) In this study, the validated Korean version questionnaire will be used
Patient Global Impression of Change (PGIC) | Finish survey by August 2020
  PGIC is an indicator that evaluates the improvement of patients in 7 steps, and the subject responds with improvement of functional limitation after treatment with 7 likert. (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).
Spine surgery | Finish survey by August 2020
  The number of spinal surgery after discharge
Current symptoms | Finish survey by August 2020
  Possible walking time without pain, neurological claudication
Treatment after discharge | Finish survey by August 2020
  Treatment history in the last month
hanbangchilyo manjogdo 9/5000 Satisfaction with integrative Korean medicine | Finish survey by August 2020
  Preference for integrative Korean medicine, satisfaction with integrative Korean medicine, How helpful hospitalization has been for returning to work and adjusting to daily life.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Dr., Study Director — Jaseng Medical Foundation
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Blood E, Hanscom B, Herkowitz H, Cammisa F, Albert T, Boden SD, Hilibrand A, Goldberg H, Berven S, An H; SPORT Investigators. Surgical versus nonsurgical therapy for lumbar spinal stenosis. N Engl J Med. 2008 Feb 21;358(8):794-810. doi: 10.1056/NEJMoa0707136. PMID 18287602
- [Background] Kalichman L, Cole R, Kim DH, Li L, Suri P, Guermazi A, Hunter DJ. Spinal stenosis prevalence and association with symptoms: the Framingham Study. Spine J. 2009 Jul;9(7):545-50. doi: 10.1016/j.spinee.2009.03.005. Epub 2009 Apr 23. PMID 19398386
- [Background] Deyo RA, Mirza SK, Martin BI. Error in trends, major medical complications, and charges associated with surgery for lumbar spinal stenosis in older adults. JAMA. 2011 Sep 14;306(10):1088. doi: 10.1001/jama.2011.1300. No abstract available. PMID 21917578
- [Background] Weinstein JN, Lurie JD, Olson PR, Bronner KK, Fisher ES. United States' trends and regional variations in lumbar spine surgery: 1992-2003. Spine (Phila Pa 1976). 2006 Nov 1;31(23):2707-14. doi: 10.1097/01.brs.0000248132.15231.fe. PMID 17077740
- [Background] Atlas SJ, Keller RB, Wu YA, Deyo RA, Singer DE. Long-term outcomes of surgical and nonsurgical management of lumbar spinal stenosis: 8 to 10 year results from the maine lumbar spine study. Spine (Phila Pa 1976). 2005 Apr 15;30(8):936-43. doi: 10.1097/01.brs.0000158953.57966.c0. PMID 15834339
- [Background] Delitto A, Piva SR, Moore CG, Welch WC. Surgery Versus Nonsurgical Treatment of Lumbar Spinal Stenosis. Ann Intern Med. 2015 Sep 1;163(5):397-8. doi: 10.7326/L15-5129-4. No abstract available. PMID 26322703
- [Background] Patel J, Osburn I, Wanaselja A, Nobles R. Optimal treatment for lumbar spinal stenosis: an update. Curr Opin Anaesthesiol. 2017 Oct;30(5):598-603. doi: 10.1097/ACO.0000000000000495. PMID 28696946
- [Background] Bodeker G. Lessons on integration from the developing world's experience. BMJ. 2001 Jan 20;322(7279):164-7. doi: 10.1136/bmj.322.7279.164. No abstract available. PMID 11159579
- [Background] Jung B, Bae S, Kim S. Use of Western Medicine and Traditional Korean Medicine for Joint Disorders: A Retrospective Comparative Analysis Based on Korean Nationwide Insurance Data. Evid Based Complement Alternat Med. 2017;2017:2038095. doi: 10.1155/2017/2038095. Epub 2017 Dec 6. PMID 29456569
- [Background] Lee YJ, Shin JS, Lee J, Kim MR, Ahn YJ, Shin YS, Park KB, Shin BC, Lee MS, Kim JH, Cho JH, Ha IH. Survey of integrative lumbar spinal stenosis treatment in Korean medicine doctors: preliminary data for clinical practice guidelines. BMC Complement Altern Med. 2017 Aug 29;17(1):425. doi: 10.1186/s12906-017-1942-6. PMID 28851418
- [Background] Hadianfard MJ, Aminlari A, Daneshian A, Safarpour AR. Effect of Acupuncture on Pain and Quality of Life in Patients with Lumbar Spinal Stenosis: A Case Series Study. J Acupunct Meridian Stud. 2016 Aug;9(4):178-82. doi: 10.1016/j.jams.2015.11.032. Epub 2015 Nov 17. PMID 27555222
- [Background] Kim K, Jeong Y, Youn Y, Choi J, Kim J, Chung W, Kim TH. Nonoperative Korean Medicine Combination Therapy for Lumbar Spinal Stenosis: A Retrospective Case-Series Study. Evid Based Complement Alternat Med. 2015;2015:263898. doi: 10.1155/2015/263898. Epub 2015 Oct 12. PMID 26543486
- [Background] Oka H, Matsudaira K, Takano Y, Kasuya D, Niiya M, Tonosu J, Fukushima M, Oshima Y, Fujii T, Tanaka S, Inanami H. A comparative study of three conservative treatments in patients with lumbar spinal stenosis: lumbar spinal stenosis with acupuncture and physical therapy study (LAP study). BMC Complement Altern Med. 2018 Jan 19;18(1):19. doi: 10.1186/s12906-018-2087-y. PMID 29351748
- [Background] Qin Z, Ding Y, Xu C, Kwong JSW, Ji Y, Wu A, Wu J, Liu Z. Acupuncture vs Noninsertive Sham Acupuncture in Aging Patients with Degenerative Lumbar Spinal Stenosis: A Randomized Controlled Trial. Am J Med. 2020 Apr;133(4):500-507.e20. doi: 10.1016/j.amjmed.2019.08.038. Epub 2019 Sep 13. PMID 31525334
- [Background] Kim KH, Kim YR, Baik SK, Noh SH, Kim DH, Lee SW, Yang GY. Acupuncture for patients with lumbar spinal stenosis: a randomised pilot trial. Acupunct Med. 2016 Aug;34(4):267-74. doi: 10.1136/acupmed-2015-010962. Epub 2016 Mar 7. PMID 26953235
- [Background] Kim KH, Kim TH, Lee BR, Kim JK, Son DW, Lee SW, Yang GY. Acupuncture for lumbar spinal stenosis: a systematic review and meta-analysis. Complement Ther Med. 2013 Oct;21(5):535-56. doi: 10.1016/j.ctim.2013.08.007. Epub 2013 Aug 20. PMID 24050593
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Jeon CH, Kim DJ, Kim SK, Kim DJ, Lee HM, Park HJ. Validation in the cross-cultural adaptation of the Korean version of the Oswestry Disability Index. J Korean Med Sci. 2006 Dec;21(6):1092-7. doi: 10.3346/jkms.2006.21.6.1092. PMID 17179693
- [Background] Kim SH, Ahn J, Ock M, Shin S, Park J, Luo N, Jo MW. The EQ-5D-5L valuation study in Korea. Qual Life Res. 2016 Jul;25(7):1845-52. doi: 10.1007/s11136-015-1205-2. Epub 2016 Mar 10. PMID 26961008
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359